CLINICAL TRIAL: NCT01415791
Title: Oral Mucosal Absorption of ICI176,334-1 in Japanese Healthy Male Subjects
Brief Title: Oral Mucosal Absorption of ICI176,334-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6874L00026
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: oral mucosal absorption; pharmacokinetics; safety; bicalutamide; Japanese; healthy subject

ARMS (1):
- Active 1 (Experimental): 8 subjects will receive ICI176,334-1
  Interventions: Drug: ICI176,334-1

INTERVENTIONS:
Drug: ICI176,334-1 — Subject will receive single dose of ICI176,334-1

SUMMARY:
The purpose of this study is to investigate the presence or absence of oral mucosal absorption of ICI176,334-1

DETAILED DESCRIPTION:
Oral mucosal absorption of ICI176,334-1 in Japanese healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Japanese healthy male subjects aged 20 to 45 years
* Male subjects should be willing to use barrier contraception ie, condoms, until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 17 and 27 kg/m2
* Eligible based on the physical findings, supine BP, pulse rate, ECG and laboratory assessments, as judged by the investigator(s)

Exclusion Criteria:

* Presence of any disease under medical treatment
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunological, blood, endocrine, neurological or mental disease to interfere with absorption, distribution, metabolism or excretion of drugs judged by investigator(s)
* Presence of any infectious disease, such as bacteria, virus and fungus Presence of allergic disorder, such as asthma, pollen disease or atopic dermatitis, and judged as necessary any medical treatment
* Any large surgical history of gastrointestinal tract such as gastric/intestinal resection or suturation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in plasma | Samples are taken at 72 hours after application of the investigational drug
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in plasma | Samples are taken at 168 hours after application of the investigational drug
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in saliva | Samples are taken at 72 hours after application of the investigational drug
To investigate the presence or absence of oral mucosal absorption of ICI176,334-1 by assessment of concentration of bicalutamide in saliva | Samples are taken at 168 hours after application of the investigational drug

SECONDARY OUTCOMES:
To assess the safety by assessment of adverse event | Adverse Events will be captured starting from screening up to 14 to 21 days (follow-up)
To evaluate the safety by evaluation of vital signs | Collect prior to treatment and up to 14 to 21 days (follow-up) after application of the investigational drug
To evaluate the safety by assessment of electrocardiograms (ECGs) | Collect prior to treatment and up to 14 to 21 days (follow-up) after application of the investigational drug